CLINICAL TRIAL: NCT01296126
Title: Structural and Functional Neuroimaging Studies of Combat Veterans
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110090; 11-N-0090
Record Dates: First submitted 2011-02-12; First posted 2011-02-15 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-02-03

CONDITIONS: Traumatic Brain Injury; PTSD
Keywords: Post Traumatic Stress Disorder (PTSD); MRI; TBI; Traumatic Brain Injury; Post Traumatic Stress Disorder; PTSD
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Studies have shown that some people develop post-traumatic stress disorder (PTSD) after being exposed to the trauma of military combat. They may have repeated thoughts, images, and dreams of the trauma; feel detached from others; have difficulty sleeping and concentrating; or be easily startled. Some studies have also shown that after having a blow or blast to the head, some people may develop post-concussive syndrome (PCS), which may include symptoms such as headaches, difficulty concentrating, and feeling moody or irritable. Researchers are interested in using magnetic resonance imaging (MRI) to study combat veterans from Operation Iraqi Freedom or Operation Enduring Freedom in order to evaluate possible changes in the brain that may be attributed to PTSD or PCS.

Objectives:

- To evaluate changes in brain function in recent combat veterans that may be related to post-traumatic stress disorder or post-concussive syndrome.

Eligibility:

- Combat veterans of Operation Iraqi Freedom/Operation Enduring Freedom who are enrolled in Walter Reed Army Medical Center protocol 351030, have returned within the last 6 weeks from a deployment in Iraq or Afghanistan that lasted at least 3 months, and are able to have magnetic resonance imaging scans.

Design:

* This study involves between 1 and 4 outpatient visits to the NIH Clinical Center over the course of 1 year. The second, third, and fourth visits will occur 3, 6, and 12 months after the first visit.
* At the first visit, participants will have a baseline MRI scan, followed by a functional MRI (fMRI) scan to see what parts of the brain are used while performing simple tasks and responding to images. Participants will complete questionnaires after the scan to report on their experiences during the MRI scan.
* For the remaining three study visits, participants will have further MRI and fMRI scans and will complete additional questionnaires. Participation is complete after the 12-month study visit, or following a diagnosis of PTSD, major depression, or PCS at any time during the study.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
Objective: Traumatic brain injury (TBI) and posttraumatic stress disorder (PTSD) are linked with functional impairments, poor outcomes compared to matched controls or people without brain dysfunction, and greater healthcare utilization. TBI can be diagnosed at the point of injury, but post-concussive syndrome (PCS) and PTSD are diagnosed after the initial exposure. Current treatments are often ineffective, and many affected military service members (SMs) never return to active duty. Upon return from deployment, many SMs experience an initial honeymoon period during which symptoms are limited in number and scope, but this may be followed by a sharp increase in symptoms within months. Identification of independent predictors of PTSD and PCS upon return from deployment could facilitate early intervention to prevent disability. The main purpose of this protocol is to determine whether structural and functional neuroimaging in SMs who are ostensibly healthy upon return can differentiate those who will go on to have persistent neurocognitive difficulties from those who will not.

Study population: The study population will be returning SMs at risk for PCS or PTSD. It involves a prospective cohort study of 128 healthy active duty military SMs, recruited by the Walter Reed National Military Medical Center (WRNMMC) from National Capital Area military units within 8 weeks after return from Iraq or Afghanistan, with serial evaluations to identify both those who develop PTSD or PCS, as well as factors obtained at the time of the initial evaluation that prove to be most strongly associated with subsequent PTSD and PCS. A comprehensive baseline assessment will be performed at WRNMMC under protocol 351030 (already approved at both the Uniformed Services University of Health Sciences [USUHS] and WRNMMC), which will include demographics, neuropsychological assessment, genetic and neuroendocrine assays, brain imaging and synchronization, vestibular, olfactory, and psychophysiologic measures. Neuroimaging and fMRI activation tasks will be performed under this imaging protocol at NIH. The study is funded by the USUHS Center for Neuroscience and Regenerative Medicine (CNRM) and NIH. See the attached WRNMMC protocol 351030.

Design: Neuroimaging including structural and functional magnetic resonance imaging (fMRI), and diffusion tension imaging (DTI) will be performed under this imaging protocol at NIH. Follow-up visits at 3, 6, and 12 months will allow repeated MRIs and fMRI activation tasks. Data analysis will include serial univariate and multivariate analyses to identify the baseline measures (including not only the results from this imaging study at NIH but also the results from a variety of studies to be performed at WRNMMC) that are most strongly associated with the subsequent development of PTSD and PCS.

Outcome measures: The primary outcome of interest is the development of neurocognitive difficulties (PCS, PTSD, or depression). Multivariate analyses will assess what baseline measures are most strongly associated with this outcome.

ELIGIBILITY:
* INCLUSION CRITERIA:

Warfighters who:

1. Are enrolled in WRNMMC protocol 351030.
2. Have returned within the previous 8 weeks from a deployment of at least 3 months duration in Iraq or Afghanistan.

EXCLUSION CRITERIA:

Warfighters who:

1. Are not able to hear normal conversation.
2. Do not have visual acuity correctable to 20/100 in at least one eye.
3. Have had a head injury resulting in loss of consciousness for 60 minutes or more or have a current Glasgow Coma Scale < 14.
4. Meet criteria for PTSD, major depression, or post-concussive syndrome at the time of the initial evaluation at WRNMMC. (A history of one or more of these conditions in the past is not exclusionary as long as criteria are not met at the time of evaluation).
5. Have active psychotic symptoms, or active suicidal or homicidal ideation, identified on the medical history, Patient Health Questionnaire, or Clinician-Administered PTSD Scale.
6. Are pregnant as shown by a pregnancy test taken during the baseline intake at WRNMMC.
7. Have retained metal fragments (shrapnel), body piercings that cannot be removed, or other imbedded ferromagnetic metal resulting from trauma or surgery, which would pose a risk for MRI scanning.
8. Have significant claustrophobia, including but not limited to intolerance of magnetic resonance imaging in the past, as we cannot provide sedating medications with the scans due to the potential impact of the medications on interpretation of scan results.
9. Report that they regularly drink 3 or more alcoholic beverages a day.
10. Report that they take illegal drugs.
11. Report that they are unable to abstain from the use of alcohol, narcotics, benzodiazepines, or sleep medication for 24 hours before being scanned.
12. Are on calcium channel blockers (e.g., verapamil, nifedipine) or alpha-blockers (e.g., prazosin, terazosin) and are unable to stop these medications for a 24-hour period prior to scanning. They will be excluded due to the impact of these medications on the interpretation of fMRI imaging.
13. Are ill with active Acinetobacter or other clinically significant infection as identified during their military evaluation upon their return from theater.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-01-26; Study Completion 2014-02-03

PRIMARY OUTCOMES:
Images from Magnetic Resonance Imaging, including structural, functional and DTI scans
Results from the cognitive neuroscience experiments

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Belliveau JW, Kennedy DN Jr, McKinstry RC, Buchbinder BR, Weisskoff RM, Cohen MS, Vevea JM, Brady TJ, Rosen BR. Functional mapping of the human visual cortex by magnetic resonance imaging. Science. 1991 Nov 1;254(5032):716-9. doi: 10.1126/science.1948051.
- [Background] Belliveau JW, Rosen BR, Kantor HL, Rzedzian RR, Kennedy DN, McKinstry RC, Vevea JM, Cohen MS, Pykett IL, Brady TJ. Functional cerebral imaging by susceptibility-contrast NMR. Magn Reson Med. 1990 Jun;14(3):538-46. doi: 10.1002/mrm.1910140311. PMID 2355835
- [Background] Blair KS, Smith BW, Mitchell DG, Morton J, Vythilingam M, Pessoa L, Fridberg D, Zametkin A, Sturman D, Nelson EE, Drevets WC, Pine DS, Martin A, Blair RJ. Modulation of emotion by cognition and cognition by emotion. Neuroimage. 2007 Mar;35(1):430-40. doi: 10.1016/j.neuroimage.2006.11.048. Epub 2007 Jan 18. PMID 17239620
- [Derived] White SF, Costanzo ME, Thornton LC, Mobley AM, Blair JR, Roy MJ. Increased cognitive control and reduced emotional interference is associated with reduced PTSD symptom severity in a trauma-exposed sample: A preliminary longitudinal study. Psychiatry Res Neuroimaging. 2018 Aug 30;278:7-12. doi: 10.1016/j.pscychresns.2018.06.006. Epub 2018 Jun 12. PMID 29935441
- [Derived] White SF, Costanzo ME, Blair JR, Roy MJ. PTSD symptom severity is associated with increased recruitment of top-down attentional control in a trauma-exposed sample. Neuroimage Clin. 2014 Nov 18;7:19-27. doi: 10.1016/j.nicl.2014.11.012. eCollection 2015. PMID 25610763